CLINICAL TRIAL: NCT04341038
Title: Open Randomized Single Centre Clinical Trial to Evaluate Methylprednisolone Pulses and Tacrolimus in Patients With Severe Lung Injury Secondary to COVID-19
Brief Title: Clinical Trial to Evaluate Methylprednisolone Pulses and Tacrolimus in Patients With COVID-19 Lung Injury
Acronym: TACROVID
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Xavier Solanich, Xavier Solanich, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TACRO-BELL-COVID; 2020-001445-39 (EudraCT Number)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Lung Injury
MeSH Terms: conditions — COVID-19; Lung Injury | interventions — Tacrolimus; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician who will finally carry out the analyses will be blind to the treatment received by the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Methylprednisolone pulses 120mg/day for 3 consecutive days (if they were not previously administered) with Tacrolimus at the necessary dose to achieve plasma levels of 8-10 ng/ml.
  In addition, these patients can receive all the treatments considered necessary for their clinical management.
  Interventions: Drug: Tacrolimus; Drug: Methylprednisolone
- Usual care (No Intervention): These patients can receive all the treatments considered necessary for their clinical management, except cyclosporine and tacrolimus.

INTERVENTIONS:
Drug: Tacrolimus — the necessary dose to obtain blood levels of 8-10 ng / ml
  Other Names: Advagraf®, Modigraf®
  Arms: Intervention
Drug: Methylprednisolone — 120mg of methylprednisolone daily for 3 consecutive days
  Other Names: Urbason®, Solu-Moderín®
  Arms: Intervention

SUMMARY:
The primary objective of the study is to evaluate the days until reaching clinical stability after starting randomization in hospitalized patients with elevated inflammatory parameters and severe COVID-19 lung injury.

DETAILED DESCRIPTION:
Unfortunately, the treatment of COVID-19 disease is still based on life support therapies. Nowadays, there is no scientific evidence from clinical trials regarding the efficacy or safety of different drugs to treat COVID-19 patients, despite some of them evolving to fatal severe lung injury due to important inflammatory process secondary to pro-inflammatory cytokines. Interestingly, Tacrolimus has been shown to inhibit both pro-inflammatory cytokines and, also, human coronavirus SARS-Cov replication, but it has not specifically been tested in COVID-19 patients.

Our working hypothesis is that severe SARS-CoV-2 (COVID-19) pneumonia is secondary to a deleterious inflammatory process; so, the use of Methylprednisolone pulses and Tacrolimus in hospitalized severe COVID-19 lung injury patients might have a positive clinical effect.

Given the COVID-19 current health emergency, this study could provide useful evidence to treat some COVID-19 patients with Methylprednisolona and Tacrolimus, which might represent a new therapeutic option for them. Tacrolimus is a drug with more than 20 years of experience, and therefore, its side effects are well known and usually reversible. In addition, since tacrolimus is a low-cost and easy to produce at large-scale drug, it could be used to treat a large number of patients. The administration of this drugs could not only decrease mortality secondary to lung involvement by COVID-19, but also decrease the excessive burden of care that intensive care units are bearing.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection confirmed by PCR
* New onset radiological infiltrates
* Respiratory failure (PaO2 / FiO2 <300 or satO2 / FiO2 <220)
* PCR>100 mg/L and/or D-Dimer>1000 µg/L and/or Ferritin>1000 ug/L
* Informed consent.

Exclusion Criteria:

* Life expectancy ≤ 24h
* Glomerular filtration ≤ 30 ml / min / 1.73 m2
* Leukopenia ≤ 4000 cells / µL
* Concomitant potentially serious infections.
* Contraindication for the use of tacrolimus according to the specifications of the product
* Known adverse reactions to treatment
* Have participated in a clinical trial in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to reach clinical stability | 28 days
  Assess the days until clinical stability is achieved after initiating randomization in hospitalized patients with elevated inflammatory parameters and severe COVID-19 lung injury.
  Clinical stability is defined if all the following criteria are met for 48 consecutive hours: Body temperature ≤ 37.0ºC; PaO2 / FiO2> 400 and / or SatO2 / FiO2> 300; Respiratory rate ≤ 24 rpm

SECONDARY OUTCOMES:
Time to reach an afebrile state for 48 hours. | 56 days
  days
Time to reach PaO2 / FiO2> 400 and / or SatO2 / FiO2> 300 | 56 days
  days
Time to reach FR ≤ 24 rpm for 48 hours | 56 days
  days
Time to normalization of D-dimer (<250 ug / L) | 56 days
  days
Time until PCR normalization (<5mg / L). | 56 days
  days
Time until normalization of ferritin (<400ug / L) | 56 days
  days
Study the impact of immunosuppressive treatment on viral load using quantitative PCR | 56 days
  viral load
Time until hospital discharge | 56 days
  days
Need for ventilatory support devices | 56 days
  days
Duration that it is necessary to maintain ventilatory support. | 56 days
  days
COVID-19 mortality | 56 days
  days
all-cause mortality | 56 days
  days
Analyze the expanded cytokine profile before the start of treatment and their evolution every 7 days after admission | 56 days
  cytokines quantification technique by Luminex
Describe the side effects and their severity attributed to tacrolimus and / or methylprednisolone. | 56 days
  IDIBELL Clinical Research and Clinical Trials Unit will oversee the monitoring and pharmacovigilance

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Corbella, MD, PhD, Study Director — Hospital Universitari de Bellvige
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solanich X, Antoli A, Rocamora-Blanch G, Padulles N, Fanlo-Maresma M, Iriarte A, Mitjavila F, Capdevila O, Riera-Mestre A, Bas J, Vicens-Zygmunt V, Niubo J, Calvo N, Bolivar S, Rigo-Bonnin R, Mensa-Vilaro A, Arregui L, Tebe C, Videla S, Hereu P, Corbella X. Methylprednisolone Pulses Plus Tacrolimus in Addition to Standard of Care vs. Standard of Care Alone in Patients With Severe COVID-19. A Randomized Controlled Trial. Front Med (Lausanne). 2021 Jun 14;8:691712. doi: 10.3389/fmed.2021.691712. eCollection 2021. PMID 34195214
- [Derived] Solanich X, Antoli A, Padulles N, Fanlo-Maresma M, Iriarte A, Mitjavila F, Capdevila O, Molina M, Sabater J, Bas J, Mensa-Vilaro A, Niubo J, Calvo N, Bolivar S, Rigo-Bonnin R, Arregui L, Tebe C, Hereu P, Videla S, Corbella X. Pragmatic, open-label, single-center, randomized, phase II clinical trial to evaluate the efficacy and safety of methylprednisolone pulses and tacrolimus in patients with severe pneumonia secondary to COVID-19: The TACROVID trial protocol. Contemp Clin Trials Commun. 2021 Mar;21:100716. doi: 10.1016/j.conctc.2021.100716. Epub 2021 Jan 19. PMID 33495742